CLINICAL TRIAL: NCT05935800
Title: The Effect of the COVID-19 Pandemic on Frailty in Liver Transplant Candidates
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 012.HEP.2022.D
Record Dates: First submitted 2023-07-06; First posted 2023-07-07 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Frailty; Sarcopenia; COVID-19
MeSH Terms: conditions — Frailty; Sarcopenia; COVID-19 | interventions — Desmoglein 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: COVID Patients who Underwent pre-transplant frailty assessment (PFA) at MDMC — This is a single-center, retrospective study that uses de-identified, anonymized patient data. Data from 369 liver transplant candidates who underwent pre-transplant frailty assessments at the Liver Institute at Methodist Dallas from April 1, 2018 to February 28, 2022. The study data will be divided into cohorts: pre-COVID and COVID. Specifically, the pre-COVID period will consist of the dates between April 1st, 2018 and March 12, 2020, while the COVID period will consist of the dates between March 13, 2020 and February 28th, 2022.

SUMMARY:
Frailty is associated with higher rates of morbidity, mortality, and failure to rescue after major surgical procedures [1]. Sarcopenia is degenerative loss of skeletal muscle mass and strength. It is a key component of physical frailty and is associated with poorer post-surgical outcomes due to decreased patient strength and vitality.

DETAILED DESCRIPTION:
This study seeks to examine whether the SARS-CoV-2 (COVID-19) pandemic, an ongoing global health crisis that was declared a national emergency by the US Federal Government on March 13, 2020, has exacerbated both frailty and sarcopenia in a population of liver transplant candidates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older Underwent pre-transplant frailty assessment (PFA) at MDMC

Exclusion Criteria:

* Not a patient at Liver Institute at Methodist Dallas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 18 years and older Underwent pre-transplant frailty assessment (PFA) at MDMC 369 liver transplant candidates who underwent pre-transplant frailty assessments at the Liver Institute at Methodist Dallas from April 1, 2018 to February 28, 2022. The study data will be divided into cohorts: pre-COVID and COVID. Specifically, the pre-COVID period will consist of the dates between April 1st, 2018 and March 12, 2020, while the COVID period will consist of the dates between March 13, 2020 and February 28th, 2022.
Sampling Method: Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of the COVID-19 pandemic on the prevalence of sarcopenia | 2 years
  To determine the impact of the COVID-19 pandemic on the prevalence of sarcopenia and frailty in patients undergoing liver transplant evaluation at Methodist Dallas Medical Center
To determine the impact of the COVID-19 pandemic on the incidence of sarcopenia | 2 years
  To determine the impact of the COVID-19 pandemic on the incidence of sarcopenia and frailty in patients undergoing liver transplant evaluation at Methodist Dallas Medical Center

SECONDARY OUTCOMES:
Changes in number of comorbidities between pre- and during/post-pandemic periods | 1 year
  Changes in number of comorbidities between pre- and during/post-pandemic periods
Changes in type of comorbidities between pre- and during/post-pandemic periods | 1 year
  Changes in type of comorbidities between pre- and during/post-pandemic periods
Changes in severity of comorbidities between pre- and during/post-pandemic periods | 1 year
  Changes in severity of comorbidities between pre- and during/post-pandemic periods

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States